CLINICAL TRIAL: NCT06224712
Title: Arogya Sangama: 3 Way Partnership of People, Providers, and Panchayat for Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Karnataka Health Promotion Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00023305
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Health Care Utilization; Health Care Seeking Behavior; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Patient Acceptance of Health Care; Behavior

STUDY DESIGN:
Intervention Model Description: The study team will use a 2 arm(intervention and control), pre and post, mixed-methods quasi experimental design comparing the intervention to the standard interventions in the area. It will be implemented in two PHC-HWCs in the Devadurga and Kollegal blocks of Raichur and Chamrajanagar districts; Two additional PHC- HWCs from these blocks similar in characteristics as the intervention PHC-HWCs will be identified as control.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arogya Sangama Intervention (Experimental): The villages in the service area of both the intervention and control PHC-HWCs will be selected randomly, weighted by population size (PPS). There are two different population groups that are being examined to get a comprehensive picture of primary health services.
  Group 1: To assess the impact of the intervention in improving the coverage and utilisation of antenatal and post-natal services, a cross-sectional sample of 1680 women, 840 in each arm, in the age group of 18-49 years who delivered in the last 12 months will be interviewed in the baseline and similarly in the endline.
  Group 2: To estimate the effect of the intervention on improving the access to screening and management of NCDs among diabetic and hypertensives, a cross-sectional sample of 200 persons in the age group of 30 years and above from each arm will be interviewed in the baseline and similarly in the endline. Hence in each round the total sample will be 400.
  Interventions: Behavioral: Arogya Sangama
- Control (No Intervention): Same inclusion criteria as above, without Arogya Sangama intervention.

INTERVENTIONS:
Behavioral: Arogya Sangama — Using human-centered design, the investigators will work wit the community to develop a prototype Arogya Sangama model to identify methods to bring GPTF and HWC service providers to create ideas, systems, processes, services, and delivery strategies for the GPTFs. They will help identify and prioritize interventions and address barriers to usability. There will also be capacity building of GPTFs to implement the interventions identified.
  Arms: Arogya Sangama Intervention

SUMMARY:
This is a two-year pilot project in the Raichur and Chamarajanagar districts of Karnataka, India aiming to enhance the overall performance of primary health systems, including service utilization, quality, and responsive care, specifically within the recently developed facilities called the Health and Wellness Centres (HWCs). It will leverage rural local government structures known as Gram Panchayat Task Forces (GPTFs) created during the Covid-19 pandemic to strengthen the services delivered by HWCs. The aim is to build capacities and empower these GPTFs to function as a collaborative platform involving people, panchayats, and healthcare providers. This approach seeks to promote-community ownership, grassroots synergy, and social accountability to strengthen HWC service delivery in rural Karnataka (India).

DETAILED DESCRIPTION:
Specific research questions:

1. What are attitudes, perceptions, and experiences of stakeholders about GPTFs involvement in the COVID 19 management and PHC service delivery?
2. What strategies and actions can GPTF undertake to improve community engagement, service provider support, and promote equitable access to essential PHC services?
3. What capacity building inputs, mechanisms, and resources will be required for GPTFs to strengthen community engagement and serve as collaborative platforms to increase social accountability for PHC services?
4. What has been the experience of GPTFs, community and program administrators about the Arogya Sangama model in terms of its applicability, adoption, and feasibility in the project settings?
5. How have GPTF interventions within Arogya Sangama project impacted community engagement, service provider support, and equitable access to essential PHC services.
6. What has been the effect of the GPTF intervention on utilization, and coverage of essential primary care services?

Empowered people and communities are a key pillar of primary health care (PHC). Within India, several policies, especially decentralization efforts under the National Health Mission had envisioned engagement of Panchayats or local self governments as a key mechanism to achieve large-scale community participation and ensure equitable access for vulnerable people, particularly women, children, and the poor. Empowering village panchayats to implement and provide oversight for National Health Ministry programs through village health committees and panchayat assemblies was expected to facilitate the process. The National Health Policy 2017 recommended an enhanced role of panchayats in health governance, including the social determinants of health and mandating community led accountability mechanisms for health to be driven by these local bodies.

States were expected to develop strategic plans and accountability mechanisms with active involvement of local self-governments for effective monitoring of quality of health care services. Despite several policies and promising vision, there is limited capacity and lack of a clear strategy for panchayat engagement and community ownership for HWCs at the state and district levels. Progress on implementing preventive and promotive services involving community and panchayats has been slow especially in aspirational districts and tribal settings. A recent evaluation of HWCs across 18 states in India including Karnataka further confirms lack of community participation as a key barrier in strengthening comprehensive primary health care (CPHC) delivery. These findings suggest a need to enable the state government to develop a clear community engagement strategy and build capacities of the panchayats in leading these efforts in the HWC service areas.

Building on the legacy of GPTF involvement in COVID 19 mitigation efforts so far, the Department of Rural Development and Panchayat Raj, (DoRDPR), within the Government of Karnataka, is proposing to strengthen and equip GPTFs with the necessary skills and tools to transform into effective forums for local health action and convergence to enhance PHC delivery. The DoRDPR has commissioned a two-year implementation research project in collaboration with the Johns Hopkins Bloomberg School of Public Health and the Karnataka Health Promotion Trust (KHPT), a leading Non Governmental Organization for Public Health action in Karnataka. The pilot project aims to build capacities of GPTFs to function as a "3-way partnership platform" (comprising of people, panchayats, and service providers) to increase community ownership, grassroots convergence, and social accountability for rural HWCs in Karnataka in Devadurga and Kollegal Block of Raichur and Chamarajanagar district respectively.

The Johns Hopkins team will use its expertise in global health and design thinking to develop interventions for GPTF based on end users' perspectives. The team, with KHPT support, will gather insights on stakeholders' perspectives about GPTF, potential new ideas, and intervention strategies required to develop GPTF as an effective 3-way partnership platform. It will develop, implement, test a prototype model, and investigate its applicability, adoption, and feasibility. It will document changes in service provision and formulate an operational framework for GPTF-enabled responsive PHC.

ELIGIBILITY:
Group 1 Inclusion criteria

* 18-49 years of age women who delivered in the last 12 months
* Residents of the districts and living within the service área covered by intervention and control PHC-HWCs
* Kannada speaking
* Able to provide consent

Group 2 inclusion criteria

* 30 or more years of age
* Not a known case of diabetes and hypertension
* Residents of the districts and living within the service area covered by intervention and control PHC-HWCs
* Kannada speaking
* Able to provide consent

Exclusion Criteria:

* Group 1: women not in the age group 18-49 years of age
* Group 2: participants younger than 30 years
* Not residing in the service area covered by intervention and control PHC-HWCs
* Unable to speak in Kannada
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4160 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of antenatal care utilization rates | 21 months
  The study team will analyze whether there is a difference in antenatal care utilization rates. The percent of early antenatal care registration (within first trimester of pregnancy) will be assessed.
Percent of non-communicable disease screening rate | 21 months
  For Group 2, the percent of non-communicable disease screenings will be assessed.
Percent of coverage of essential primary health care (PHC) services | 21 months
  The study team will analyze whether there is a difference in coverage of essential PHC services.
Percent of patients satisfied with treatment | 21 months
  The study team will analyze percent of patients satisfied with the treatment at the Health and Wellness Centres

CONTACTS AND LOCATIONS:
Overall Officials: Svea Closser, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- India (2):
  - Devadurga Block PHC-HWC, Devadurga
  - Kollegal PHC-HWC, Kollegāl

IPD SHARING:
Plan to Share IPD: No